CLINICAL TRIAL: NCT03688516
Title: Effects of Emotion on Episodic Memory in Typically Developing Children and Children With Williams-Beuren Syndrome
Acronym: EEM-TAdev
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2017-A03321-52
Record Dates: First submitted 2018-07-02; First posted 2018-09-28 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Mental Disorders
Keywords: emotion; memory; Williams-Beuren syndrome
MeSH Terms: conditions — Mental Disorders; Williams Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atypical development (Experimental): 30 children with Williams-Beuren syndrome will be presented with two tasks of episodic memory, one with visual stimuli and another one with audio-verbal stimuli. Manipulation of valence and modality (negative, positive, neutral) in order to measure influence of emotion on episodic memory:Spatial and recognition memory ans source and content memory. The tasks will be presented one after another with a break of 15 minutes. In both tasks the participants will have to encode the stimuli and then first recall them and second to recognize the encoded stimuli amongst new stimuli. The stimuli will be presented on the computer. The responses will be collected by the experimenter for recall task and by the computer for recognition task. During the recognition task the EEG recording will be done.
  Interventions: Behavioral: Manipulation of valence and modality; Behavioral: Spatial and recognition memory; Behavioral: Source and content memory
- Typical development (Sham Comparator): 30 control children matched for mental age will be presented with two tasks of episodic memory, one with visual stimuli and another one with audio-verbal stimuli. Manipulation of valence and modality (negative, positive, neutral) in order to measure influence of emotion on episodic memory:Spatial and recognition memory ans source and content memory. The tasks will be presented one after another with a break of 15 minutes. In both tasks the participants will have to encode the stimuli and then first recall them and second to recognize the encoded stimuli amongst new stimuli. The stimuli will be presented on the computer. The responses will be collected by the experimenter for recall task and by the computer for recognition task. During the recognition task the EEG recording will be done.
  Interventions: Behavioral: Manipulation of valence and modality; Behavioral: Spatial and recognition memory; Behavioral: Source and content memory

INTERVENTIONS:
Behavioral: Manipulation of valence and modality — mnemic task with a phase of encoding negative, positive and neutral stimuli, will be proposed followed by an immediate recovery phase, composed of a recall task followed by a recognition task
Behavioral: Spatial and recognition memory — mnemic task with a phase of encoding negative, positive and neutral stimuli, will be proposed followed by an immediate recovery phase, composed of a recall task followed by a recognition task
Behavioral: Source and content memory — mnemic task with a phase of encoding negative, positive and neutral stimuli, will be proposed followed by an immediate recovery phase, composed of a recall task followed by a recognition task

SUMMARY:
It's well established in the literature that emotional events are more likely to be remembered than neutral events. Although this Emotional Enhancement of Memory (EEM) has been well demonstrated in the adult literature, little is known about EEM for typically developing children and children with Williams-Beuren syndrome (WBS). In this study, two investigations will be conducted concomitantly: one of EEM in typically developing children and the other of EEM in children with WBS. For this purpose, three behavioral experiments will be established to investigate EEM in this two populations, with the first experiment also including electroencephalography measures. Performances of typically developing children will be compared to young adults, and performances of children with WBS will be compared to control children matched for mental age. Finally, this study aims to bring new knowledge about the interactions between emotion and memory in children, and to better understand cognitive functioning in children with WBS.

DETAILED DESCRIPTION:
The main objective of the present project is to characterize the emotional modulation of episodic memory in typically developing (TD) children and children with Williams-Beuren syndrome (WBS), by using behavioral and encephalography (EEG) measures. Better understanding of interaction between cognition and emotion in TD children and in WBS, and their specificities may increase our knowledge of normal and pathological neurodevelopment and lead to new treatment strategies in a case of WBS. Indeed, it is worth to note that WBS have a strong impact on cognitive, emotional and social aspects of children's behavior in daily life. It was widely shown in animal and human studies that emotionally charged information is better memorized and retrieved than neutral one.This emotional enhancement of memory (EEM) was largely demonstrated with young and older adults independently of the nature of stimuli, the type of memory, the type of memory task and the delay between encoding and retrieval . There is general agreement about emotional regulation of memory in adults, although there are several points currently investigated.

Surprisingly, less is known about EEM in TD children and neurodevelopmental disorders such as WBS. Availability of cognitive resources and emotional regulation is supposed to have an impact on EEM. As both present specific patterns in TD children as compared to adults and in children with WBS , it could be expected that emotional regulation of memory process in TD children and WB presents also some specificities. These specificities are largely unknown, moreover if one considers that neither memory function nor emotional processing are fully developed in TD children.

Few studies that investigated EEM in TD children reported rather contradictory results. Some of them observed EEM and others did not.In addition, most studies used only negative stimuli. Even less is known about EEM in children presenting neurodevelopmental pathologies as WBS, although memory deficit for non-emotional stimuli and deficit in processing of facial expressions, especially negative ones were observed in children with WBS. In addition, a significant dissociation was documented in children with WBS, concerning memory deficit, with auditive-verbal memory rather speared and visuo-spatial memory rather impaired .

Thus, there is an important shortcoming in our understanding of emotional modulation of memory in children, both typically developing and those presenting WBS. With the present project, the investigators propose to fill this gap: two investigations will be conducted concomitantly, one of EEM in typically developing children and the other of EEM in children with WBS. Three behavioral experiments will be established to investigate EEM in this two populations, with the first experiment also including electroencephalography measures. These experiments will address the following specific questions: (1) is the EEM dependent of the stimulus type (images versus words)? - Experiment 1; (2) does the EEM exist in visuospatial episodic memory? - Experiment 2; (3) does the EEM exist for content and source memory - Experiment 3. Performance of typically developing children will be compared to young adults, and performance of children with WBS will be compared to control children matched for mental age.

ELIGIBILITY:
Inclusion Criteria:

Children with William-Beuren syndrome

* Genetic diagnosis (CGH-Array or FISH) of microdeletion 7q11.23
* 8 to 18 years old
* Native French speaker
* Psychotropic medication unchanged during one month preceding inclusion

Typically developing children and healthy adults:

* 6 to 30 years old
* Native French speaker
* Absence of history of neurodevelopmental neurological and psychiatric disease

Exclusion Criteria:

Children with William-Beuren syndrome:

* Diagnosis of severe intellectual deficit (Total IQ lower than 40 evaluated with WPPSI-II or WISC-IV)
* Presence of another genetic anomaly
* Presence of vascular; infectious or neurodegenerative disease
* Medication impacting motor and cognitive abilities
* Non-corrected visual and hearing impairment

Typically developing children and Healthy Adults :

* Diagnosis of severe intellectual deficit (Total IQ lower than 70 evaluated with WPPSI-II or WISC-IV)
* Presence of vascular; infectious or neurodegenerative disease knew by parents or legal representative
* Learning disorders
* History of neurological or psychiatric disease
* Medication impacting motor and cognitive abilities, non-corrected visual and hearing impairment

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Manipulation of Valence | During the presentation of the stimuli or just after the presentation of the stimuli
  Behavioral measure:number of correct responses (correct recall and correct recognition), evoked potential for EEG only for Experiment 1

SECONDARY OUTCOMES:
EEG measures | During the presentation of the stimuli or just after the presentation of the stimuli
  Number of correct responses (correct recall and correct recognition), evoked potential for EEG only for Experiment 1
Source memory | During the presentation of the stimuli or just after the presentation of the stimuli
  Number of correct responses (correct recall and correct recognition), evoked potential for EEG only for Experiment 1
Content memory | During the presentation of the stimuli or just after the presentation of the stimuli
  Number of correct responses (correct recall and correct recognition), evoked potential for EEG only for Experiment 1
Spatial memory | During the presentation of the stimuli or just after the presentation of the stimuli
  Behavioral measure:number of correct responses (correct recall and correct recognition), evoked potential for EEG only for Experiment 1
Recognition memory | During the presentation of the stimuli or just after the presentation of the stimuli
  Behavioral measure:number of correct responses (correct recall and correct recognition), evoked potential for EEG only for Experiment 1
Modality of Valence | During the presentation of the stimuli or just after the presentation of the stimuli
  Behavioral measure:number of correct responses (correct recall and correct recognition), evoked potential for EEG only for Experiment 1

CONTACTS AND LOCATIONS:
Overall Officials: DEMILY CAROLINE, Principal Investigator — CH LE VINATIER
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No